CLINICAL TRIAL: NCT05635266
Title: A Single-Site Tissue Repository Providing Annotated Biospecimens for Approved Investigator-directed Biomedical Research Initiatives
Brief Title: Tissue Repository Providing Annotated Biospecimens for Approved Investigator-directed Biomedical Research Initiatives
Status: Recruiting | Type: Observational
Sponsor: Sanguine Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: SAN-BB-02
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Age-Related Macular Degeneration; Allergies; Alpha-Gal Syndrome; Alzheimer Disease; Amyloidosis; Ankylosing Spondylitis; Arthritis; Alopecia Areata; Asthma; Atopic Dermatitis; Autism; Autoimmune Hepatitis; Behcet's Disease; Beta-Thalassemia; Cancer; Celiac Disease; Kidney Diseases; COPD; Crohn Disease; Cystic Fibrosis; Diabetes; Dravet Syndrome; DMD; Fibromyalgia; Graves Disease; Thyroid Diseases; Hepatitis; Hidradenitis Suppurativa; ITP; Leukemia; ALS; Lupus or SLE; Lymphoma; Multiple Sclerosis; Myasthenia Gravis; Heart Diseases; Parkinson Disease; Pemphigus Vulgaris; Cirrhosis; Psoriasis; Schizophrenia; Scleroderma; Sickle Cell Disease; Stroke; Ulcerative Colitis; Vasculitis; Vitiligo
MeSH Terms: conditions — Macular Degeneration; Hypersensitivity; red meat allergy; Alzheimer Disease; Amyloidosis; Spondylitis, Ankylosing; Arthritis; Alopecia Areata; Asthma; Dermatitis, Atopic; Autistic Disorder; Hepatitis, Autoimmune; Behcet Syndrome; beta-Thalassemia; Neoplasms; Celiac Disease; Kidney Diseases; Pulmonary Disease, Chronic Obstructive; Crohn Disease; Cystic Fibrosis; Diabetes Mellitus; Epilepsies, Myoclonic; Fibromyalgia; Graves Disease; Thyroid Diseases; Hepatitis; Hidradenitis Suppurativa; Leukemia; Lupus Erythematosus, Systemic; Lymphoma; Multiple Sclerosis; Myasthenia Gravis; Heart Diseases; Parkinson Disease; Pemphigus; Fibrosis; Psoriasis; Schizophrenia; Scleroderma, Diffuse; Anemia, Sickle Cell; Stroke; Colitis, Ulcerative; Vasculitis; Vitiligo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Health Condition Group
  Interventions: Diagnostic Test: Specimen sample
- Exceptive Condition Group
  Interventions: Diagnostic Test: Specimen sample
- Control Group
  Interventions: Diagnostic Test: Specimen sample

INTERVENTIONS:
Diagnostic Test: Specimen sample — The study may require a tissue collection and/or a participant survey for participation. Most tissue collected will come from a blood draw; up to 100mL for the health condition group, 60mL for the exceptive condition group, and up to 180mL for the control group (if determined safe for the participant). Participant surveys may involve participant reported outcomes (PROs) or custom participant surveys.

SUMMARY:
To collect, preserve, and/or distribute annotated biospecimens and associated medical data to institutionally approved, investigator-directed biomedical research to discover and develop new treatments, diagnostics, and preventative methods for specific and complex conditions.

ELIGIBILITY:
Inclusion Criteria:

* Persons 18 to 85 years of age at the date of informed consent.
* If presenting with a history of a specific condition, the diagnosis is confirmable in the medical record or may be confirmed using other forms of verification including self-reporting.
* Understands the procedures and requirements of the study by providing written informed consent (or verbal assent if a legally authorized representative will sign the ICF), including consent for authorization for protected health information disclosure.

Exclusion Criteria:

* Persons younger than 18 years of age or older than 85 years of age at the date of informed consent.
* Receipt of blood products 30 days before the study blood draw.
* Receipt of an investigational (unapproved) drug 30 days before the study blood draw.
* A confirmable diagnosis of any medical condition that would increase potential phlebotomy risks.
* Has donated a unit of blood within the last 2 months at the date of informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health condition, exceptive condition, and control participants will be recruited by one or any of the following resources, but not limited to:
  * Use of online marketing where potential participants receive study information from the Sanguine's website or online participant referral program;
  * In the site investigators (or PI's) clinic; and/or
  * Through community advocacy programs.
  * Participant Referral
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Biospecimen & Clinical Data Collection | 10 years
  To collect enough biospecimens and associated clinical data to allow researchers to come to statistically relevant scientific results

CONTACTS AND LOCATIONS:
Overall Officials: Houman Hemmati, MD, Principal Investigator — Sanguine Biosciences
Locations (1):
- Sanguine Biosciences, Waltham, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol (2021-12-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT05635266/Prot_000.pdf